CLINICAL TRIAL: NCT05137366
Title: Transthoracic Ultrasound Evaluation of Thoracic Aortic Aneurysms
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RHMCAR0603
Record Dates: First submitted 2021-11-16; First posted 2021-11-30 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Thoracic Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Thoracic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Known Thoracic aortic aneurysm (TAA): * A medical confirmed TAA defined as an aneurysm measuring >3cm in the thoracic aorta e.g. aortic arch, ascending aorta or descending thoracic aorta.
  * Patients may also have a AAA
  * Patients may have had a TEVAR and will have a residual sac
  * A CT scan of the aorta in the last 3 years
  Interventions: Diagnostic Test: Transthoracic ultrasound scan
- Control group: A medically diagnosed Abdominal aortic aneurysm with a CT scan showing no TAA in the last three years. Patients who have also had their AAA repaired will also be eligible for this group.
  Interventions: Diagnostic Test: Transthoracic ultrasound scan

INTERVENTIONS:
Diagnostic Test: Transthoracic ultrasound scan — An ultrasound scan of the thoracic aorta will be performed using an ultrasound machine with 2 MHz phased array transducer. The patient will lay supine on an ultrasound scan couch.The measurements will be taken in B-mode but colour Doppler imaging may be used to identify the thoracic aorta if it is obscured by artefacts. The measurement will be taken inner wall to inner wall and several images will be taken to check reliability.
  Three different acoustic windows will be used to image the thoracic aorta:
  1. Suprasternal window
  2. Parasternal long axis window
  3. Apical two chamber views
  Ultrasound assessment will be considered satisfactory when at least two of the three regions of the descending thoracic aorta were visualised, partially satisfactory when a single view was obtained and inconclusive when none of the three windows could be obtained.

SUMMARY:
The Diagnosis of a thoracic Aortic Aneruysms usually made when imaging an abdominal aortic aneurysm which has reached threshold or as an incidental finding during a chest scan by computed tomography (CT) or magnetic resonance imaging (MRI). However, these imaging modalities are expensive, involve radiation exposure and can cause anaphylaxis and other allergic reaction from the contract agents used. In addition CT scans are contraindicated for those who have: allergic reactions to the contrast, radioactive iodine treatment for thyroid disease, metformin use, and chronic or acutely worsening renal disease.

Ultrasound is a non-invasive imaging modality that is cheaper than the methods currently used for TAA detection and surveillance. Echocardiography is limited in assessing the TAA as it is not sensitive to image beyond the proximal ascending aorta which is why it is currently not used for screening or surveillance.

A pilot study found that ultrasound has the potential to be used as a diagnostic modality for thoracic aortic aneurysms and may have a role in surveillance in patients for whom CT scanning is contraindicated. They found that the sensitivity and specificity of detecting TAA was 100% and 70% for a threshold of 35 mm, and 84% and 90% for a threshold of 40 mm. However, further validation of this methodology is required for it to be considered as a method of diagnosis and surveillance for this patient group. This study was only carried out by one experienced sonographer so it important to repeat this study to see if other sonographers are able to obtain the necessary views.

The main purpose of this study is to validate the protocol used by pilot study to assess whether thoracic aortic aneurysms can be detected and measured accurately using ultrasound.

There are two main objectives of this study:

1. Can ultrasound be used to detect thoracic aortic aneurysms?
2. Can ultrasound be used to accurately measure thoracic aortic aneurysms?

If the results of this study show that ultrasound has high sensitivity and specificity for detecting thoracic aortic aneurysms, it could lead to a thoracic aorta screening programme.

DETAILED DESCRIPTION:
It is important to state that patients involved in this study will not have any changes made to their routine care as a result of this study. All patients recruited would have had a recent CT scan which will be used for the comparison and will not be exposed to any additional radiation as part of the study. The CT scan used will be from the last 3 years so no new diagnoses are expected as a result of the study.

Patients There will be two different groups recruited for this study; Group 1- patients with known thoracic aortic aneurysm (TAA) and Group 2- patients with known abdominal aortic aneurysm (AAA) but no thoracic aortic aneurysm. The known TAA group will be obtained from those who are currently having CT surveillance for either a known TAA or TEVAR (Thoracic Endovascular Repair). The known AAA but no TAA will be obtained from patients who are either under for CT surveillance AAA or EVAR (Endovascular Aneurysm Repair). All patients recruited for this study will be under CT surveillance at Southampton General Hospital or Queen Alexandra hospital and would have had a CT scan within the last 3 years at University Hospital Southampton so no new findings would be expected to come from the study. In addition, the CT scan used will be part of their routine care and there will be no change to their routine care or surveillance as a result of this study.

Both Males and Female participants will be recruited for the study and there will also be a minimum age of 18 as gender will not influence the results of the study.

Participant Recruitment Any patients eligible for the study will be contacted to see if they are interested in taking part and given a participant information sheet. The participant information sheet (PIS) will entail the full details of the study and what it will involve for the patient.

If a patient is interested in participating in the study, a telephone call appointment will be arranged between a member of the research team and the patient. This phone call will involve going through the PIS, answering any questions, and obtaining verbal informed consent. During this appointment, an ultrasound scan appointment will also be arranged.

A referral for the scan will be placed by Ben Patterson using the hospitals e-quest system under the patients hospital number so that images can be stored and a report can be generated and recorded for the patients record. The referral will placed using the code UAOTD and when the referral is on the CRIS system, one of the researchers will insure that the patient is changed to a research scan to ensure that it does not interfere with routine care.

At the ultrasound assessment, written informed consent will be obtained prior to the scan being carried out and there will also be another opportunity for patients to ask any questions. If patients' are unable to consent to the study themselves as they are deemed to have a lack of capacity, they will not be included within the research study and will continue with their routine care.

Collection of demographic data Patients age and gender will be recorded for the study. No other demographic information will be recorded.

Ultrasound scan protocol A single vascular sonographer (Hannah Davey) will complete all ultrasound scans for this study and will be blinded to the CT diagnosis, location, and extent of the aortic pathology in all patients. This will be achieved by a member of the research team arranging the patients' appointment and having a study participant code for the scan referral so that the different groups cannot be identified. The vascular sonographer will also not complete any of the consenting in order to ensure they are blinded to any patient identifiable information.

The maximum diameter (inner wall to inner wall) of the different areas of the thoracic aorta will be measured; primarily focusing on the descending thoracic aorta from the isthmus to the level of the diaphragm will be obtained and recorded for the study. The sensitivity and specificity of detecting TAA will be test at measurements of both 35mm and 40mm

All scans of the thoracic aorta will be performed using a Philips Epiq 5 or Epiq 7 machine with 2 MHz phased array transducer. The patient will lay supine on an ultrasound scan couch which can be tilted in order to optimise the patient position and views required for the scan. The measurements will be taken in B-mode but colour Doppler imaging may be used to identify the thoracic aorta if it is obscured by artefacts. The measurement will be taken inner wall to inner wall and several images will be taken to check reliability.

Three different acoustic windows will be used to image the thoracic aorta:

1. Suprasternal window- To visualise aortic arch and the three major supra-aortic vessels
2. Parasternal long axis window- To visualise the mid descending thoracic aorta
3. Apical two chamber views- To visualise the distal end of the thoracic aorta and proximal segment of the abdominal aorta Ultrasound assessment will be considered satisfactory when at least two of the three regions of the descending thoracic aorta were visualised, partially satisfactory when a single view was obtained and inconclusive when none of the three windows could be obtained The ultrasound scan appointment is estimated to take approximately 30 mins for obtaining written informed consent and completing the scan. All images and measurements taken during the scan will be stored on PACS and a report for the scan will be written on CRIS.

CT Scan protocol

A consultant vascular surgeon (Mr B Patterson) at Southampton General Hospital will review the CT scans and measure the maximum diameter (inner wall to inner wall) of the thoracic aorta. He is highly experienced in imaging patients with thoracic aortic pathology so the measurements will be reliable and valid. All CT scan measurements will be carried out on the picture archiving systems (PACS) at Southampton General Hospital and will also be compared to the measurement reported on system. Similarly to the ultrasound protocol, the maximum diameter of the different areas of the thoracic aorta will be obtained and recorded for the study. The diameter used for the study will be measured inner wall to inner wall in order to allow for comparison and accuracy to the ultrasound scan.

The CT scan used for the measurement will be taken from the most recent aorta scan on the CRIS and PACS systems at Southampton General Hospital or Queen Alexandra Hospital. Patients will not be having any additional scans as part of this study and measurements will only be used from scans as part of their routine care. This is in order to minimise the amount of radiation each patient is exposed too and to make sure that their routine care is not interrupted by them participating in this study.

Images from both the ultrasound scan and CT scan will be stored on a Picture archiving and communication system (PACS). Measurements of the maximum diameter for the ultrasound scan will be completed at the time scan and will be done using the measurement software in the ultrasound machine. The CT scan measurements will be carried out on the PACS system and will be compared to the value reported in the original report to check the accuracy.

Measurements from both the ultrasound and CT scan will be recorded on Microsoft Excel. For each group, mean and standard deviation will be calculated. The sensitivity and specificity of the ultrasound scan will be analysed using cut-off points of both 35mm and 40mm. This will be done using the CT scan measurement as a reference for comparing the accuracy of the ultrasound measurement. Statistical analysis will be carried out on Statistical Package for the Social Sciences (SPSS).

In order to calculate the sensitivity and specificity of ultrasound, a Clopper-Pearson confidence interval will be carried out on Statistical Package for the Social Sciences (SPSS). The statistical analysis will be completed with a 95% confidence interval and will be calculated at both 35mm and 40mm cut-offs.

ELIGIBILITY:
Inclusion Criteria:

* For both the Thoracic Aortic Aneurysm (TAA) group and control group, there are no exclusion criteria for gender, ethnicity or socioeconomic status. However, all patients must have a minimum age of 18 years. Patients must have a diagnosis of a Thoracic Aortic Aneurysm or/and Abdominal aortic aneurysm (AAA)

The Thoracic Aortic Aneurysm groups will have:

* A medical confirmed TAA defined as an aneurysm measuring >3cm in the thoracic aorta e.g. aortic arch, ascending aorta or descending thoracic aorta.
* Patients may also have a AAA
* Patients may have had a TEVAR and will have a residual sac
* A CT scan of the aorta in the last 3 years

The Abdominal aortic aneurysm A medically diagnosed Abdominal aortic aneurysm with a CT scan showing no TAA in the last three years. Patients who have also had their AAA repaired will also be eligible for this group.

Exclusion Criteria:

* • No diagnosed TAA or AAA

  * No CT scan of aorta in last 3 years
  * Under 18 years old
  * Patient who are unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients recruited will be under the care of the Wessex vascular network at Southampton General Hospital. All patients will be identified using a key work search on CT scans from the last 5 years. This will be carried out by a member of the radiology research team at Southampton General Hospital.
  Participants who would be eligible for the TAA group would be identified by completing a keyword search of reports on the radiology information system (CRIS). The search will look for any CT scans with the following key words:
  * Thoracic aorta
  * Thoracic aortic aneurysm
  * TAAA
  * TEVAR
  * Ectatic Thoracic Aorta
  Participants who would be eligible for the AAA group with no known TAA would also be identified by completing a keyword search of reports on CRIS. The search will look for any CT scans with the following key words:
  * Abdominal aorta
  * Abdominal aortic aneurysm
  * AAA
  * EVAR
  * Ectatic abdominal Aorta
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-04-11 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Can ultrasound detect thoracic aortic aneurysms | 6 months
  Specificity and sensitivity of ultrasound in detecting thoracic aortic aneurysms
Can thoracic aortic aneurysms be accurately measured using ultrasound | 6 months
  Specificity and sensitivity of ultrasound in measuring thoracic aortic aneurysms

CONTACTS AND LOCATIONS:
Overall Officials: Ben Patterson, Principal Investigator — University Hospital Southampton NHS Foundation Trust
Locations (1):
- Southampton General Hospital, Southampton, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Access to the final study database will on be allowed for the main researchers of the study and the co-investigators listed on the participant information sheet. The data will be stored on a secure radiology drive on the trust computer system.
  Archiving will be authorised by the Sponsor following submission of the end of study report.
  Location and duration of record retention for:
  * Essential documents: Patient case notes will be stored and maintained according to standard rules and procedures. Pathology results are stored and maintained according to standard procedures.
  * Study data will be held for minimum of 5 years